CLINICAL TRIAL: NCT04175067
Title: Assessment of Thiol Disulfide Balance in Early Stage Endometrium Cancer
Brief Title: Evaluation of Thiol Disulfide Balance in Stage 1 Endometrium Cancer
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Burak Sezgin, Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: 09/08/2018-13-9
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Endometrium Cancer; Oxidative Stress
Keywords: Early stage; thiol disulfide hemostasis; malignancy
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum blood samples for aech participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometrium cancer: stage I endometrium cancer n=57
  Interventions: Diagnostic Test: Disulphide(μmol/L); Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L)
- Healthy controls: Healthy volunteers n=60
  Interventions: Diagnostic Test: Disulphide(μmol/L); Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L)

INTERVENTIONS:
Diagnostic Test: Disulphide(μmol/L) — Aforementioned oxidative stress markers will be measured via Cobas c501(Roche Diagnostics, Indianapolis, IN, USA) used with sphectrophotometry
  Other Names: Native thiol (μmol/L); Total thiol (μmol/L); Nativethiol/totalthiol(%); Disulfide/nativethiol(%); Disulfide/totalthiol(%)
Diagnostic Test: Total Oxidant Capacity(μmolH2O2Equiv/L) — Aforementioned oxidative stress markers will be measured via Cobas c501(Roche Diagnostics, Indianapolis, IN, USA) used with sphectrophotometry
  Other Names: Total Antioxidant Capacity(mmolTroloxEquiv/L); Oxidative stress Index (Arbitrary Unite)

SUMMARY:
The purpose of this study is to investigate thiol-disulfide balance in early stage endometrium cancer patients.

DETAILED DESCRIPTION:
To date various oxidative stress paramaters were studied in patients with endometrial cancer, however dynamic thiol disulfide hemostasis has not been previously investigated.

The thiol-disulfide balance in the circulation will be measured by the automated system created by Erel & Neselioglu(1).

References

1- Erel O, Neselioglu S. A novel and automated assay for thiol/disulphide homeostasis. Clin Biochem 2014;47:326-32. doi:10.1016/j.clinbiochem.2014.09.026.

ELIGIBILITY:
Inclusion Criteria:

• Histopathologically confirmed diagnosis of stage I endometrium cancer

Exclusion Criteria:

* pulmonary disease
* pulmonary hypertension
* cardiac dysfunction
* renal dysfunction
* liver disease
* chronic ishemia
* systemic inflammation
* concomitant malignancy
* patients who use vitamin A,C or E (antioxidant vitamins)
* patients who use smoke
* patients who use drink alcohol
* patients who use addictive for any drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — endometrium cancer
Study Population: The preoperative diagnosis of Endometrium cancer was made histopathologically by endometrial biopsy. An experienced pathologist performed frozen section analysis according to the surgical staging scheme of the International Federation of Gynaecology and Obstetrics.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
serum native thiol level | preoperative in the morning or preprandial for healthy volunteers
  serum native thiol level in μmol/L
serum disulphide level | preoperative in the morning or preprandial for healthy volunteers
  serum disulphide level in μmol/L
serum total thiol level | preoperative in the morning or preprandial for healthy volunteers
  serum total thiol level in μmol/L
the disulphide/native thiol ratio | preoperative in the morning or preprandial for healthy volunteers
  the disulphide/native thiol ratio X (100 )
disulphide/total thiol ratio | preoperative in the morning or preprandial for healthy volunteers
  disulphide/total thiol ratio X (100 )
native thiol/total thiol ratio | preoperative in the morning or preprandial for healthy volunteers
  native thiol/total thiol ratio X (100 )

SECONDARY OUTCOMES:
total antioxidant capacity (TAC) | preoperative in the morning or preprandial for healthy volunteers
  TAC in mmol trolox equivalent/L
total oxidant capacity (TOC) | preoperative in the morning or preprandial for healthy volunteers
  TOC in mmol H2O2 equivalent/L.
Oxidative stress index (OSI) | preoperative in the morning or preprandial for healthy volunteers
  OSI in mmol trolox/L.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Sezgin, Principal Investigator — Mugla Sıtkı Kocman University Faculty of Medicine
Locations (1):
- Mugla Sıtkı Kocman University Faculty of Medicine, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided